CLINICAL TRIAL: NCT03202225
Title: Primary Constrained Condylar Knee Arthroplasty Without Stem Extensions: Prevalence and Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Other Study IDs: COA 61/2560
Record Dates: First submitted 2017-06-25; First posted 2017-06-28 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-11

CONDITIONS: Constrained Insert in Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: constrained polyethylene — constrained polyethylene insert

SUMMARY:
While performing a primary TKA in consecutive patients, a constrained insert may be necessary when adequate stability and soft tissue balance are not obtained. In this retrospective study, The investigators aim to identify the prevalence and risk factors that associate with the use of a constrained insert in primary TKA.

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis
* primary total knee replacement

Exclusion Criteria:

* secondary knee osteoarthritis
* revision total knee replacement
* previous knee surgery
* post-traumatic knee
* history of previously infection
* comorbidity;rheumatoid arthritis, connective tissue disease, neuromuscular disease, lumbar spinal stenosis, neuropathy
* severe osteoporosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients underwent primary total knee arthroplasty at our institution
Sampling Method: Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
prevalence to use constrained insert in primary total knee arthroplasty | intraoperative
  to identify the prevalence that associate with the use of a constrained insert in primary total knee arthroplasty
risk factors to use constrained insert in primary total knee arthroplasty | intraoperative
  to identify the risk factors that associate with the use of a constrained insert in primary total knee arthroplasty such as degree of preoperative deformity, degree of preoperative instability

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — Department of Orthopaedics, Faculty of Medicine Vajira Hospital, Navamindradhiraj University
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No